CLINICAL TRIAL: NCT00673348
Title: A Prospective Observational Study of Plasma Voriconazole Concentration Measurement and Its Correlation With CYP2C19 Genotype in Korean Patients
Brief Title: Therapeutic Drug Monitoring (TDM) of Voriconazole and Correlation With CYP2C19 Genotype in Korean Populations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Dong-Gun Lee / Assistant Professor, Division of Infectious Diseases, Department of Internal Medicine
Other Study IDs: VCZ_TDM_Korea
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-06

CONDITIONS: Mycoses; Neutropenia; Bone Marrow Transplantation
Keywords: Mycoses; Voriconazole
MeSH Terms: conditions — Mycoses; Neutropenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Two times of venous blood sampling will be carried out at steady state. Three ml of venous blood is sampled right before the morning dose (trough sampling). The second sampling is carried out at any time point within 2-4 hours after the morning dose (peak sampling). To obtain the exact dose and sampling history, at least three dosing times around the trough and peak sampling will be recorded to the minute. Sampling time will also be recorded as clock time.
  * Genotyping of CYP2C19 will also be performed using 3 ml of peripheral blood sampled into EDTA tubes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients suspected of invasive fungal infection (proven or probable cases) with immunocompromised state (for example, during neutropenia, receiving HSCT) in Catholic Hematopoietic Stem Cell Transplantation [HSCT] Center in Seoul, Korea.

SUMMARY:
Voriconazole (VCZ), the antifungal drug active against Candida and Aspergillus is a substrate of CYP2C19, whose proportion of poor metabolizers is about ~20% in Asian population. The AUC's of VCZ differs over 4 folds by CYP2C19 genotypes of homozygotic wild type, heterozygote, and homozygotic poor metabolizers. The Asian population enrolled in the metabolism of VCZ were mainly Japanese and Chinese, without Korean subjects. The proportion of poor metabolizers in Korean population is known to be around 12% (Pharmacogenetics. 1996 Dec;6(6):547-51). The importance of CYP2C19 genotypes on the pharmacokinetics (PK) of voriconazole is well established, Hence, it is desirable to individualize the dosage regimen of VCZ according to the genotypes of patients. Fungal infection in immunocompromised patients is a life threatening condition which needs critical care. Although the PK change by genotypes are well known, its clinical implication or need for different dosage regimen by genotypes is not established, yet.

DETAILED DESCRIPTION:
The investigators are trying to set up voriconazole (VCZ) therapeutic drug monitoring (TDM) & establish relationship with efficacy and safety in Korea. The investigators also want to propose the optimal dosage regimen for VCZ over different genotypes of CYP2C19 in the immunocompromised patients in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised adults who are treated with voriconazole due to proven or probable invasive fungal infections

Exclusion Criteria:

* Patients who have been treated with other investigational drugs
* Patients with liver dysfunction (aminotransferase level ≥ 5 times the upper limit of normal, bilirubin or alkaline phosphatase level > 3 times the upper limit of normal)
* Patients with renal dysfunction (Cr level > 2.5 times the upper limit of normal)
* Pregnant women
* Patients younger than 15 years of age

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of invasive fungal infection (proven or probable cases) with immunocompromised state (for example, during neutropenia, receiving HSCT) in Catholic Hematopoietic Stem Cell Transplantation [HSCT] Center in Seoul, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To regular setting of voriconazole TDM & establish relationship with efficacy and safety | Prospective

SECONDARY OUTCOMES:
To apply population pharmacokinetic-pharmacodynamic modeling and simulation technique on the clinical research of antifungal drugs. | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Gun Lee, M.D., Ph.D., Principal Investigator — St. Mary's Hospital, The Catholic Univ. of Korea
Locations (1):
- St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim SH, Yim DS, Choi SM, Kwon JC, Han S, Lee DG, Park C, Kwon EY, Park SH, Choi JH, Yoo JH. Voriconazole-related severe adverse events: clinical application of therapeutic drug monitoring in Korean patients. Int J Infect Dis. 2011 Nov;15(11):e753-8. doi: 10.1016/j.ijid.2011.06.004. Epub 2011 Aug 9. PMID 21831685